CLINICAL TRIAL: NCT05443126
Title: A Modular, Open-label, Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of EP0031 in Patients With Advanced RET-altered Malignancies
Brief Title: A Study of EP0031 in Patients With Advanced RET-altered Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ellipses Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP0031-101
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; NSCLC
Keywords: selective RET-inhibitor; NSCLC; RET

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- RET fusion-positive NSCLC (prior 1st gen SRI) (Experimental): EP0031 capsules at the recommended phII dose, taken once daily until progressive disease (PD), unacceptable toxicity or patient withdrawal
  Interventions: Drug: EP0031
- RET mutation-positive MTC (prior 1st gen SRI) (Experimental): EP0031 capsules at the recommended phII dose, taken once daily until progressive disease (PD), unacceptable toxicity or patient withdrawal
  Interventions: Drug: EP0031
- Other RET-altered solid tumours (prior 1st gen SRI) (Experimental): EP0031 capsules at the recommended phII dose, taken once daily until progressive disease (PD), unacceptable toxicity or patient withdrawal
  Interventions: Drug: EP0031
- RET fusion-positive NSCLC (no prior SRI therapy) (Experimental): EP0031 capsules at the recommended phII dose, taken once daily until progressive disease (PD), unacceptable toxicity or patient withdrawal
  Interventions: Drug: EP0031
- RET mutation-positive MTC (no prior SRI therapy) (Experimental): EP0031 capsules at the recommended phII dose, taken once daily until progressive disease (PD), unacceptable toxicity or patient withdrawal
  Interventions: Drug: EP0031
- Other RET-altered solid tumours (no prior SRI therapy) (Experimental): EP0031 capsules at the recommended phII dose, taken once daily until progressive disease (PD), unacceptable toxicity or patient withdrawal
  Interventions: Drug: EP0031

INTERVENTIONS:
Drug: EP0031 — EP0031 is a potent next-generation selective RET-inhibitor (SRI)

SUMMARY:
The aim of this study is to assess the safety, side effects and effectiveness of EP0031 in patients with advanced RET-altered malignancies (NSCLC)

DETAILED DESCRIPTION:
EP0031 is being investigated in this modular, interventional Phase I/II dose escalation and dose expansion study to investigate the optimal dose in adult patients with advanced RET-altered malignancies. Currently there are no approved RET-targeted treatments for patients who progress on first-generation SRIs. However, it is proposed that EP0031 can overcome resistance mechanisms to first generation SRIs, as EP0031 is a potent and selective RET inhibitor with broad activity against common RET fusions and mutations. Phase I (dose escalation and optimization) has completed and a RP2D has been selected for Phase II.

ELIGIBILITY:
Inclusion Criteria:

Applicable to all patients:

1. Must be ≥18 years of age, with documented RET-altered cancers
2. Patients should be well informed and consented about alternative treatment options including approved RET-targeted therapies
3. ECOG performance status of 0 or 1 and life expectancy >3 months at screening
4. Ability to understand and provide written informed consent and able to participate in all required evaluations and procedures
5. Additional cohort specific criteria apply

Exclusion Criteria:

Patients with any of the following will not be included in the study:

1. Any known major driver gene alterations other than RET.
2. Spinal cord compression or brain metastases. Patients with stable brain metastases can be enrolled.
3. Active infection requiring systemic antibiotic, antifungal, or antiviral medication
4. Severe or uncontrolled medical condition or psychiatric condition
5. Chronic glomerulonephritis or renal transplant
6. Patients with active hepatitis B infection or active hepatitis C
7. Patients with active HIV infection. Patients living with HIV may be eligible if they have adequate CD4+ T-cell count and no history of AIDS-defining opportunistic infections in the past 12 months
8. Receipt of any strong inhibitor or inducer of CYP3A4
9. Impaired hepatic or renal function, inadequate bone marrow reserve or organ function
10. Any clinically important abnormalities in rhythm, conduction, or morphology on resting ECG or any factor that increases the risk of QTc prolongation or of arrhythmic events , or congestive heart failure Grade II-IV according to the New York Heart Association, myocardial infarction, or unstable angina within the previous 6 months
11. Uncontrolled hypertension
12. Corneal ulceration at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Module A: Incidence of Dose-limiting Toxicity (DLTs ) during the first 28 days of EP0031 treatment | First 28 days of treatment
Modules B and C: Overall Response Rate (ORR) as measured using RECIST v1.1 | 12 months

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | First 48 hours after drug administered
  To characterise the pharmacokinetics (PK) of EP0031
Maximum Plasma Concentration (Cmax) | First 24 hours after drug administered
  To characterise the pharmacokinetics (PK) of EP0031
Time taken for drug concentration to fall from half its original value (Half-life) | First 72 hours after drug administered
  To characterise the pharmacokinetics (PK) of EP0031

CONTACTS AND LOCATIONS:
Locations (40):
- United States (18):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Cancer Specialist, Fort Myers, Florida
  - RUSH University Medical Center, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYU Langone Health, New York, New York
  - Providence Portland Medical Centre, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Washington University, Seattle, Washington
  - Seattle Cancer Care / Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (5):
  - Assistance publique - Hôpitaux de Marseille, Marseille, Bouches-du-Rhône
  - Center Bergonié, Bordeaux, Gironde
  - Institut Gustave-Roussy, Villejuif, Paris
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
- Charité Comprehensive Cancer Center, Berlin, Germany
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy
- Spain (7):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
  - University Hospital October 12, Madrid
  - Hospital Madrid Sanchinarro, Madrid
  - Hospital Virgen de la Victoria de Malaga, Málaga
- United Arab Emirates (3):
  - Tawam Hospital, Al Ain City, Abu Dhabi Emirate
  - Sheik Shakhbout Medical City (SSMC), Abu Dhabi
  - Cleveland Clinic Abu Dhabi (CCAD), Abu Dhabi
- United Kingdom (5):
  - University College London Hospital, London
  - Guy's Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield